CLINICAL TRIAL: NCT05942807
Title: The Prognostic and Predictive Role of Clinical, Biochemical, Pathological and Molecular Characteristics of Patients With Biliary Tract Cancer: an Observational Monocentric Study. (BABEL)
Brief Title: Observational Monocentric Study on Biliary Tract Cancer (BABEL)
Acronym: BABEL
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 4173
Record Dates: First submitted 2023-03-20; First posted 2023-07-12 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
BABEL is an observational, single-center, prospective study about patients affected by biliary tract cancers (BTC) treated at the Medical Oncology Unit of the FPUAG - IRCCS.

DETAILED DESCRIPTION:
BABEL is an observational, single-center, prospective study with an historical cohort. Study population is represented by patients affected by biliary tract cancers (BTC) treated at the Medical Oncology Unit of the FPUAG - IRCCS. The study involves an historical cohort and a prospective cohort. Primary aim of the study is to associate BTC patients' overall survival with IDH1/2 mutations, in order to confirm the prognostic role of these genes both metastatic and resectable disease setting. The secondary aims are to correlate FGFR mutations and overall survival of BTC patients and to find new clinical and molecular characteristics linked with survival and response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biliary tract cancer;
* Patients with radiological evident disease;
* Patients >18 anni;
* Written informed consent;
* Patients with at least one oncological visit.

Exclusion Criteria:

* Patients without available clinical data;
* Patients without histological diagnosis of BTC;
* Patients without written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population is consituited by patients with BTC treated at Medical Oncology Unit of the FPUAG - IRCCS. The study involves a historical cohort and a prospective cohort.
Sampling Method: Probability Sample
Enrollment: 560 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Overall survival | The expected OS for BTC patients is 18 months
  OS is defined as the time between patient's date of diagnosis and date of death from any cause of the patient. For patients with no observed event, the follow-up time will be ended to the same date.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Salvatore, MD, PhD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (1):
- Fondazione Policlinico Universitario Agostino Gemelli/IRCSS - UOC di Oncologia Medica, Roma, Rome, Italy